CLINICAL TRIAL: NCT00216099
Title: A Phase II Study of Pemetrexed (Alimta) as Second-Line Therapy for Hormone Refractory Prostate Cancer: Hoosier Oncology Group GU03-67
Brief Title: Pemetrexed as Second-Line Therapy in Treating Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Sweeney, MBBS (Other)
Collaborators: Eli Lilly and Company (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Christopher Sweeney, MBBS, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GU03-67
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pemetrexed; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): * Pemetrexed 500 mg/m2 IV over 10 minutes, day 1 of 21-day cycle
  * Oral Folic Acid, once per day for 7 days preceding pemetrexed dose, continued daily, and for 21 days after the last dose of pemetrexed.
  * Vitamin B12, 1000ug intramuscular injection 7 days preceding pemetrexed dose, and every three cycles thereafter on the same day of pemetrexed administration
  Interventions: Drug: Pemetrexed; Dietary Supplement: Folic Acid; Dietary Supplement: Vitamin B12

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV over 10 minutes, day 1 of 21-day cycle
  Other Names: Alimta
Dietary Supplement: Folic Acid — All participants received oral Folic Acid 350-100ug once per day for 7 days preceding the first pemetrexed dose and continuing throughout the study and and for 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 — All patients received vitamin B12 1000ug intramuscular injection the week preceding the first pemetrexed dose and received additional 1000ug intramuscular injections every three cycles thereafter on the same day of pemetrexed administration.

SUMMARY:
Docetaxel-based therapy has been shown to prolong survival as first-line therapy for patients with hormone refractory prostate cancer (HRPC), and has become the standard of care. The beneficial effects of any therapy in HRPC may be diverse and include reduction in tumor bulk (when measurable), reduction in prostate-specific antigen PSA, reduction in symptoms (particularly pain), or stabilization of disease. Clear reductions in tumor bulk or PSA may provide objective evidence of a treatment effect, and stabilization of disease may be just as clinically meaningful in patients who are actively progressing prior to starting therapy. Pemetrexed has shown a broad array of activity in many diseases that until now were thought to be non-responsive to chemotherapy in the second-line setting.

This trial is designed to further assess the efficacy, safety, tolerability, and pharmacogenetics of pemetrexed as a single agent in subjects with HRPC whose disease has progressed following one prior taxane-based chemotherapy regimen for HRPC.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Pemetrexed 500mg/m2 will be administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle.
* Folic Acid (350-1000 mcg. PO daily) will be taken by patients to reduce toxicity. At least 5 daily doses of folic acid must be taken during the 7-day period preceding the first dose of pemetrexed, and dosing should continue during the full course of therapy and for 21 days after the last dose of pemetrexed.
* Vitamin B12 (1000 µg) will be administered as an intramuscular injection during the week preceding the first dose of pemetrexed and every 3 cycles thereafter. Subsequent vitamin B12 injections may be given the same day as pemetrexed.

Performance Status: Karnofsky Performance Status 70-100

Life expectancy > 12 weeks

Hematopoietic:

* Absolute Neutrophil Count (ANC) > 1500/mm3
* Platelet count > 100,000/mm3
* Hemoglobin > 9 g/dL

Hepatic:

* Bilirubin < 1.5 X upper limit of normal (unless due to Gilbert's disease)
* Alkaline phosphatase and Alanine Transanimase (ALT) (SGPT) < 3 X upper limit of normal (ULN); may be < 5 X ULN for patients with liver metastases. Alkaline phosphatase may be any value for patients with bone metastases.

Renal:

* Calculated creatinine clearance >45 mL/min based on the standard Cockroft and Gault formula

Cardiovascular:

* No congestive heart failure requiring therapy or New York Heart Association (NYHA) class II or greater or active angina or known myocardial infarction within 12 months prior to study
* No unstable angina, uncontrolled congestive heart failure, or unstable symptomatic arrhythmia requiring medication within 6 months prior to being registered for protocol therapy
* Subjects with chronic atrial arrhythmia, i.e., atrial fibrillation, paroxysmal supraventricular tachycardia, or controlled hypertension are eligible

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Clinically refractory or resistant to hormone therapy as assessed by progression following at least one hormonal therapy (orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist)
* One prior taxane based chemotherapy regimen for HRPC
* Documented progression of disease after one taxane based prior chemotherapy regimen for HRPC. Progression is defined as at least one of the following:
* An increase in PSA > 50% over nadir value on prior Taxane-based therapy
* Progression of measurable disease as defined by RECIST
* Progression of bone disease as defined by the appearance of one or more new bone lesions or worsening symptoms
* Orchiectomy or testosterone levels < 50 ng/dL maintained by LHRH agonist
* Prior chemotherapy, or other experimental anticancer agents must be completed > 4 weeks prior to being registered for protocol therapy
* Palliative radiotherapy must be completed at least 14 days prior to registration.

Exclusion Criteria:

* Intravenous radio-isotopes therapy must be completed at least 6 weeks prior to registration
* No brain metastasis that are untreated and/or not controlled and/or still requiring corticosteroids
* No history of other malignancies within 5 years prior to being registered for protocol therapy, except for adequately treated basal or squamous cell skin cancer
* No history of uncontrolled psychiatric illness or serious systemic disease, including active infection, uncontrolled hypertension
* No surgery or significant traumatic injury within 21 days prior to being registered for protocol therapy
* Patients must be willing to interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5-day period (8 day period for long acting agents such as piroxicam)
* Patients must be willing to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, M.B.B.S., Study Chair — Hoosier Oncology Group, LLC
Locations (15):
- United States (15):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Center for Hematology/Oncology of S. Michigan, Jackson, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates S.J., P.A., Mount Holly, New Jersey
  - Consultants in Medical Oncology & Hematology, Drexel Hill, Pennsylvania
  - Pennsylvania Oncology-Hematology Associates, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hahn NM, Zon RT, Yu M, Ademuyiwa FO, Jones T, Dugan W, Whalen C, Shanmugam R, Skaar T, Sweeney CJ. A phase II study of pemetrexed as second-line chemotherapy for the treatment of metastatic castrate-resistant prostate cancer (CRPC); Hoosier Oncology Group GU03-67. Ann Oncol. 2009 Dec;20(12):1971-6. doi: 10.1093/annonc/mdp244. Epub 2009 Jul 15. PMID 19605506
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed 500mg/m^2: Pemetrexed 500 mg/m2 IV over 10 minutes, day 1 of 21-day cycle
  Pemetrexed: Pemetrexed 500 mg/m2 IV over 10 minutes, day 1 of 21-day cycle
Period: Overall Study
Arm/Group | Pemetrexed 500mg/m^2
Started | 49
Toxicity Analysis | 49
Response Analysis | 48
Completed | 48
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 68 [58 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 49
Baseline Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] — Prostate-Specific Antigen (PSA) is a protein produced by the prostate in men. Elevated PSA levels (>4ng/mL) can be an indicator of infection or cancer of the prostate.
  ng/mL | 72.2 [0.8 to 1015.0]
Baseline Karnofsky Performance Status (KPS) [Median (Full Range); unit: units on a scale] — Karnofsky Performance Status (KPS) is a general indicator of a subject's well being and ability to carry on daily activities. The KPS scale ranges from 0-100 in 10 unit increments where 100=Normal; no complaints; no evidence of disease and 0=Dead
  units on a scale | 90 [70 to 100]
Baseline Pain Score [Median (Full Range); unit: units on a scale] — Patients self-scored their pain on a scale of 0-10 where 0=no pain and 10=extreme pain
  units on a scale | 2 [0 to 10]
Baseline Opiate Use [Mean (Full Range); unit: Intramuscular morphine equivalents] | 9.6 [0 to 80]
Metastatic Sites [Number; unit: participants] — Number of patients who had metastatic disease present at the specified site at trial entry
  participants
    Bone | 31
    Lymph Node | 16
    Visceral | 7
Days Since Last Docetaxel [Number; unit: participants]
  0-28 | 30
  29-90 | 7
  91-180 | 5
  >180 | 6
  unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall PSA Response
Description: Best overall Prostate-Specific Antigen (PSA) response
  PSA response is defined by a greater than or equal to 50% decline in PSA confirmed by a second PSA value at least 4 weeks after the first PSA response timepoint PSA Stable Disease is defined as less than a 50% decline in PSA and less than a 50% increase in PSA from baseline PSA progression is defined as greater than or equal to a 50% increase in PSA compared to baseline
Time Frame: Start of treatment until disease progression/recurrence (for life)
Measure: Number (95% Confidence Interval); unit: percentage of participatns
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 49
percentage of participatns
  >50% decline in PSA | 8 [1 to 16]
  Stable PSA | 20 [9 to 32]
  PSA progression | 65 [52 to 79]

2. Secondary Outcome: Overall Survival
Time Frame: From study enrollment until death (for life)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 48
months | 14 [13 to 19.0]

3. Secondary Outcome: OBJECTIVE Overall Response Rate
Description: Response Evaluation Criteria in Solid Tumors (RECIST). Objective overall response rate is defined as Complete Response (CR) + Partial Response (PR)
  Per RECIST:
  CR= Disappearance of all target and non-target lesions and normalization of tumor marker level PR= Disappearance of all target lesions and persistence of non-target lesion(s) or maintenance of tumor marker level above normal limits OR at least a 30% decrease in the sum of the longest diameter, taking as reference the baseline sum longest diameter and disappearance of all non-target lesions or persistence of non-target lesion(s) or maintenance of tumor marker level above normal limits
Time Frame: Start of treatment until disease progression/recurrence (for life)
Population: Patients who had measurable disease per RECIST 1.1 at baseline. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension with longest diameter >20 mm using conventional techniques or >10 mm with spiral CT scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 26
percentage of participants
  Participants with PR with meas. dis. per RECIST | 8 [1 to 25]
  participants with SD maintained at 12 weeks | 39 [20 to 59]

4. Secondary Outcome: Rate of Clinical Benefit
Description: A clinical benefit is defined as an improvement for at least 3 consecutive weeks in at least one of the following parameters without any sustained worsening in any other:
  > 50% reduction in analgesic consumption or > 50% reduction in pain intensity or > 20 point gain in performance status.
Time Frame: Any time among evaluable subjects (for life)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 48
percentage of participants | 33 [20 to 48]

5. Secondary Outcome: Safety and Tolerability
Description: Safety and Tolerability was evaluated by reporting the percentage of patient who experienced grade 3 or 4 toxicities using Common Terminology Criteria for Adverse Events CTCAE v3.0 criteria. CTCAE grades the severity of an adverse event from 1-5 where 1=least severe and 5=death.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 49
percentage of participants
  Grade 3 | 42.9 [27 to 55.8]
  Grade 4 | 8.2 [2.3 to 19.6]

6. Secondary Outcome: RFC1 G80A Genotype
Description: Samples for RFC1 G80A pharmacogenetic analysis were collected at screening
Time Frame: Screening
Population: Samples were available from 46 patients
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 46
participants
  A/A Genotype | 6
  A/G Genotype | 22
  G/G Genotype | 18

7. Secondary Outcome: Time to Progression
Description: Progression per Response Evaluation Criteria in Solid Tumors (RECIST) or Prostate-Specific Antigen (PSA) Progression RECIST PD=at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions PSA progression=increase in PSA to >50% above lowest level recorded on study. Two consecutive increases required at least 4 weeks apart, but time to progression will be determined at time of first PSA showing increase > 50% above baseline *Note, upper confidence interval was not reached*
Time Frame: Study enrollment until progression per RECIST or PSA (for life)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 48
months | 5 [1 to NA] — The upper confidence interval was not reached.

8. Secondary Outcome: Time to Prostate-Specific Antigen (PSA)/Serological Progression
Description: Serological Progression (sPD) - increase in PSA to >50% above lowest level recorded on study. Two consecutive increases required at least 4 weeks apart, but time to progression will be determined at time of first PSA showing increase > 50% above baseline
Time Frame: From study enrollment to progression per PSA criteria (for life)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 500mg/m^2
Number analyzed (Participants) | 48
months | 2 [1 to 5]

ADVERSE EVENTS:
Time Frame: Duration of Treatment
Arm/Group | Pemetrexed 500mg/m^2
Serious Adverse Events (participants affected / at risk) | 15/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed 500mg/m^2 (N=49)
CONFUSION (Nervous system disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DIC (DISSEMINATED INTRAVASCULAR COAGULATION) (Blood and lymphatic system disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1 (1)
FEBRILE NEUTROPENIA(ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
HEMORRHAGE, CNS (Nervous system disorders) | 1 (1)
HEPATOBILIARY/PANCREAS - OTHER (Hepatobiliary disorders) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / CATHETER-RELATED (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / SKIN (CELLULITES) (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 1 (1)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / CARDIAC/HEART (Cardiac disorders) | 1 (1)
PAIN / PELVIS (General disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 1 (1)
VESSEL INJURY-ARTERY / EXTREMITY-LOWER (Vascular disorders) | 1 (2)
VESSEL INJURY-VEIN / EXTREMITY-LOWER (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed 500mg/m^2 (N=49)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 1 (1)
ALKALINE PHOSPHATASE (Investigations) | 7 (8)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 1 (1)
ALLERGY/IMMUNOLOGY - OTHER (Immune system disorders) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 6 (7)
ANOREXIA (Gastrointestinal disorders) | 17 (32)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 2 (2)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 5 (7)
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 1 (1)
CARDIAC GENERAL - OTHER (Cardiac disorders) | 2 (2)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 10 (17)
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (15)
CREATININE (Investigations) | 7 (10)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 2 (3)
DIARRHEA (Gastrointestinal disorders) | 13 (18)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (3)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 13 (21)
EDEMA: LIMB (Blood and lymphatic system disorders) | 12 (15)
EDEMA: TRUNK/GENITAL (Blood and lymphatic system disorders) | 1 (1)
EXTRAPYRAMIDAL/INVOLUNTARY MOVEMENT/RESTLESSNESS (Nervous system disorders) | 2 (2)
EXTREMITY-LOWER (GAIT/WALKING) (Musculoskeletal and connective tissue disorders) | 3 (3)
EXTREMITY-UPPER (FUNCTION) (Musculoskeletal and connective tissue disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 41 (65)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 2 (2)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 9 (20)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 1 (1)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 3 (3)
GYNECOMASTIA (Reproductive system and breast disorders) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 9 (9)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 11 (12)
HEMOGLOBIN (Blood and lymphatic system disorders) | 21 (44)
HEMOGLOBINURIA (Investigations) | 1 (3)
HEMORRHAGE, GI (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, GI / ANUS (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES/FLUSHES (Endocrine disorders) | 6 (6)
HYPERTENSION (Cardiac disorders) | 3 (3)
HYPOTENSION (Cardiac disorders) | 1 (1)
INCONTINENCE, URINARY (Renal and urinary disorders) | 1 (1)
INFECTION - OTHER (Infections and infestations) | 5 (5)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BLADDER (URINARY) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / ABDOMEN NOS (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / BLADDER (URINARY) (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / LYMPHATIC (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / SKIN (CELLULITES) (Infections and infestations) | 1 (2)
INFECTION WITH UNKNOWN ANC / UPPER AIRWAY NOS (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 4 (8)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Surgical and medical procedures) | 1 (1)
INSOMNIA (General disorders) | 13 (15)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 4 (13)
LUMBAR SPINE-RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 1 (1)
LYMPHATICS - OTHER (Blood and lymphatic system disorders) | 1 (4)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 7 (8)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 8 (9)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 4 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Gastrointestinal disorders) | 2 (2)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 5 (5)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 3 (3)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 1 (1)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 22 (34)
NEUROLOGY - OTHER (Nervous system disorders) | 1 (1)
NEUROPATHY: MOTOR (Nervous system disorders) | 5 (5)
NEUROPATHY: SENSORY (Nervous system disorders) | 11 (12)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 3 (4)
OBSTRUCTION, GU / PROSTATE (Reproductive system and breast disorders) | 1 (1)
OCULAR/VISUAL - OTHER (Eye disorders) | 2 (3)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 3 (3)
PAIN / BACK (General disorders) | 13 (14)
PAIN / BLADDER (Renal and urinary disorders) | 1 (1)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 8 (12)
PAIN / BREAST (Reproductive system and breast disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 9 (11)
PAIN / EXTREMITY-LIMB- HAND (General disorders) | 1 (1)
PAIN / EYE (Eye disorders) | 1 (2)
PAIN / HEAD/HEADACHE (General disorders) | 2 (2)
PAIN / INTESTINE (Gastrointestinal disorders) | 1 (1)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / NEURALGIA/PERIPHERAL NERVE (Nervous system disorders) | 1 (1)
PAIN / ORAL CAVITY (Gastrointestinal disorders) | 1 (1)
PAIN / PERINEUM (General disorders) | 1 (1)
PAIN / PROSTATE (Reproductive system and breast disorders) | 1 (3)
PAIN / RECTUM (Gastrointestinal disorders) | 1 (2)
PAIN / SCALP (General disorders) | 1 (1)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1)
PAIN - OTHER (General disorders) | 5 (7)
PAIN - OTHER FEET (General disorders) | 1 (1)
PAIN / BACK (General disorders) | 2 (2)
PAIN / EXTREMITY-LIMB (General disorders) | 2 (3)
PAIN / EYE (Eye disorders) | 1 (1)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 4 (5)
PAIN / PELVIS (General disorders) | 1 (1)
PANCREATITIS (Hepatobiliary disorders) | 1 (1)
PETECHIAE/PURPURA (HEMORRHAGE/BLEEDING INTO SKIN OR MUCOSA) (Gastrointestinal disorders) | 1 (1)
PETECHIAE/PURPURA (HEMORRHAGE/BLEEDING INTO SKIN OR MUCOSA) (Vascular disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 6 (9)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 9 (11)
PTT (PARTIAL THROMBOPLASTIN TIME) (Surgical and medical procedures) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 6 (7)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 8 (13)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 3 (3)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 (1)
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 1 (1)
RIGORS/CHILLS (General disorders) | 3 (3)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 6 (8)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 4 (5)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 2 (2)
URINE COLOR CHANGE (Renal and urinary disorders) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 11 (16)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 9 (10)
WEIGHT LOSS (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No